CLINICAL TRIAL: NCT00978900
Title: Carbohydrates and Non Caloric Sweeteners: Differential Effects on Appetite and Secretion of Gastrointestinal Satiety Peptide
Brief Title: Effects of Artificial Sweetener on Gastrointestinal (GI) Peptide Secretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Beglinger Christoph, Prof. Dr. med., Department of Gastroenterology, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 69/04
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: satiety peptides; GLP-1; PYY; ghrelin; appetite profile; Sweetening Agents
MeSH Terms: interventions — Sweetening Agents; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Acesulfame K (Active Comparator)
  Interventions: Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars
- Sucralose (Active Comparator)
  Interventions: Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars
- Aspartame (Active Comparator)
  Interventions: Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars
- Glucose (Active Comparator)
  Interventions: Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars
- Fructose (Active Comparator)
  Interventions: Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars
- Water (Placebo Comparator)
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Artificial sweeteners; Carbohydrate Sugars — sweetening agent dissolved in tap water, administered via intragastric tube
  Arms: Acesulfame K; Aspartame; Fructose; Glucose; Sucralose
Dietary Supplement: Water
  Arms: Water

SUMMARY:
The purpose of this study is to examine the influence of artificial sweeteners (aspartame, acesulfame K, sucralose) and carbohydrate sugars (glucose, fructose) on the release of gastrointestinal satiety hormones in humans.

DETAILED DESCRIPTION:
Artificial Sweeteners significantly lower energy density of foods and beverages. They are used by diabetics as sugar substitutes as well as by consumers as aids for dietary control. Despite numerous studies which show mainly no influence of artificial sweeteners on glucose metabolism and food intake, discrepancies consist about the real effects of artificial sweeteners. Studies by Blundell and Hill in 1986 have however shown that the consumption of artificial sweeteners resulted in an increase of appetite ratings; the efficiency of AS has therefore been questioned. With respect to the world wide increase in the prevalence in obesity, it seems important to clarify whether artificial sweeteners can help regulate body weight or not. This study will explore the effect of artificial sweeteners on the release of the gastrointestinal satiety hormones PYY, GLP-1, GIP and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject with a body-mass index of 19.0-24.5
* Normal eating habits
* Age 18-40 years
* Stable body weight for at least three months

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medications (except for oral contraceptives)
* Medical or psychiatric illness
* history of gastrointestinal disorders
* food allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal peptide secretion | 2 hour blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Clinical Research Center, University Hospital Basel